CLINICAL TRIAL: NCT06665477
Title: A Randomized, No-treatment-controlled, Evaluator-blinded, Multi-center Study to Evaluate the Effectiveness and Safety of Restylane Volyme in the Treatment of Temple Hollowing
Brief Title: Evaluate the Effectiveness and Safety of Restylane Volyme in the Treatment of Temple Hollowing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43CH2401
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Temple Hollowing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subject treated with Restylane Volyme (Experimental)
  Interventions: Device: Restylane Volyme
- Subject non-treated with Restylane Volyme (No Intervention)

INTERVENTIONS:
Device: Restylane Volyme — Subjects in Restylane Volyme treatment group will receive treatment on Day 1 and optiponal treatment 1 month later.
  Arms: Subject treated with Restylane Volyme

SUMMARY:
A randomized, no-treatment-controlled, evaluator-blinded, multi-center study to evaluate the effectiveness and safety of Restylane Volyme in the treatment of temple hollowing

ELIGIBILITY:
Inclusion Criteria:

1. Ability to adequately understand the verbal explanations and the written subject information provided in local language and ability and willingness to give consent to participate in the study. Signed and dated informed consent to participate in the study.
2. Males or non-pregnant, non-breastfeeding females of Chinese origin and 18 years of age or older at the time of signing the Informed Consent Form (ICF).
3. Grade 2 (moderate) to 3 (severe) on the 4-grade GTVDS for both temples as assessed by the Blinded Evaluator as well as the Treating Investigator on Day 1 (agreement on grade is not required). The GTVDS grade for the right temple and the left temple does not have to be equal but must not differ by more than 1 grade.
4. Willing to abstain from any other facial plastic surgical or cosmetic procedures above the level of the horizontal line from subnasale for the duration of the study (e.g., laser or chemical resurfacing, needling, facelift, lifting threads, radiofrequency etc.).
5. Intent to undergo treatment for correction of temple hollowing.

   Inclusion criteria 6-7 apply to female subjects only:
6. If the subject is a female of childbearing potential, she agrees to use an acceptable form of effective birth control for the duration of the study and is willing to take a urine pregnancy test (UPT) or a serum HCG (blood test [if UPT is not available]) at screening, baseline and prior to receiving any study treatment.

   Acceptable forms of effective birth control include:
   * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical caps) with spermicidal foam/gel/film/cream/suppository;
   * Bilateral tubal ligation;
   * Combined oral contraceptives (estrogens and progesterone), implanted or injectable contraceptives on a stable dose for at least 28 days prior to Day 1;
   * Hormonal or copper intra uterine device (IUD) inserted at least 28 days prior to Day 1;
   * Vasectomized partner (in monogamous relationship) for at least 3 months prior to screening;
   * Strict abstinence (at least one month prior to baseline and agrees to continue for the duration of the study or use acceptable form of birth control).
7. Negative pregnancy test for women of childbearing potential at the screening and baseline visits.

Exclusion Criteria:

1. Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel or to gram positive bacterial proteins.
2. Known/previous allergy or hypersensitivity to local anesthetics, e.g., lidocaine or other amide-type anesthetics or nerve blocking agents (if intended to be used for that subject).
3. Previous or present severe or multiple allergies manifested by severe reactions, such as anaphylaxis or angioedema, or family history of these conditions.
4. Previous facial surgery (e.g., facelift) above the level of the horizontal line from subnasale that in the Treating Investigator´s opinion could interfere with the study safety and/or effectiveness assessments.
5. Any previous aesthetic procedures or implants:

   * Previous permanent filler or implant, lifting threads, or autologous fat in the face regardless of time.
   * Previous use of calcium hydroxylapatite (CaHA) or poly-L-lactic acid (PLLA) above the level of the horizontal line from subnasale within 24 months.
   * Previous HA filler or collagen filler above the level of the horizontal line from subnasale within 12 months.
   * Previous botulinum toxin treatment above the level of the horizontal line from subnasale within 6 months.
   * Previous energy based aesthetic procedures (e.g., laser, intense pulsed light, radiofrequency, photomodulation and ultrasound) above the level of the horizontal line from subnasale within 6 months.
   * Previous mechanical (e.g., dermabrasion, needling) or chemical aesthetic procedures (e.g., chemical peel) above the level of the horizontal line from subnasale within 6 months.
   * Previous treatment with cryotherapy above the level of the horizontal line from subnasale within 6 months.
6. History of cancer or previous radiation above the level of the horizontal line from subnasale.
7. Presence of any disease or lesions near or on the area to be treated, e.g.:

   * Inflammation, active or chronic infection (e.g., in mouth, dentals, head, eye);
   * Facial psoriasis, eczema, acne, rosacea, perioral dermatitis, herpes simplex or herpes zoster;
   * Scars or deformities;
   * Cancer, or precancerous conditions (e.g., actinic keratosis or actinic cheilitis).
8. Evidence of scar-related disease or delayed healing activity within 1 year prior to the baseline visit, or subjects susceptible to keloid formation, hyperpigmentation or hypertrophic scarring in the opinion of the Investigator.
9. Presence of tattoo, piercing, beard or facial hair, which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessment.
10. Recurrent temporal headaches such as temporal tendinitis migraine. Have a history of migraines or frequent headaches, as determined by the (Treating) Investigator, that could interfere with the study safety and/or effectiveness assessments.
11. History of temporomandibular joint disorder, jaw pain, chewing pain or muscular related pain in the treatment area.
12. Temple hollowing due to trauma, congenital malformations, or lipodystrophy, either congenital or acquired.
13. Experienced trauma to the temple area within 6 months before enrollment or has residual deficiencies, deformities, or scarring.
14. Temporal arteritis or history of temporal arteritis.
15. Presence of a dental, oral, or facial condition which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessments, e.g., has dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities. Any planned procedure (e.g., dental implants, tooth extractions, orthodontia) during the study period, that would make the subject unsuitable for inclusion in the opinion of the Investigator.
16. Abnormal/moderate or abnormal/severe score for temple firmness or detection of any abnormal temple structure, such as lump/mass formation or non-uniform density.
17. Abnormal/moderate or abnormal/severe score for temple symmetry.
18. An underlying known disease, a surgical or medical condition that would expose the subject to undue risk, e.g., history of bleeding disorders, active hepatitis, active autoimmune disease such as, connective tissue diseases systemic lupus erythematosus, polymyositis, dermatomyositis, or scleroderma.
19. Use of concomitant medication that have the potential to prolong bleeding times such as anticoagulants or inhibitors of platelet aggregation (e.g., direct factor Xa inhibitors, warfarin, clopidogrel, aspirin or other non-steroidal anti-inflammatory drugs [NSAIDs], Omega 3 or Vitamin E), within 14 days prior to injection. Omega 3 and Vitamin E are acceptable only as part of a standard multivitamin formulation. Cyclooxygenase-2 (COX 2) inhibitors are allowed.
20. Treatment with chemotherapy, immunosuppressive agents, systemic corticosteroids within 3 months before treatment (inhaled corticosteroids are allowed).
21. Use of topical facial corticosteroids or prescription retinoids near or on the area to be treated within 1 month of the baseline visit or systemic retinoid treatment within 6 months of the baseline visit, or plan to receive such treatment during participation in the study.
22. Presence of any condition or situation, which in the opinion of the Treating Investigator makes the subject unable to complete the study per protocol, e.g.

    * Subject is not likely to avoid other prohibited facial cosmetic treatments;
    * Subject is not likely to complete the study because of other commitments;
    * Subject is anticipated to be unavailable for visits, incapable of understanding the investigational assessments or having unrealistic expectations of treatment result;
    * Subject who has a concomitant condition (e.g., acute viral or bacterial infection with fever) that might confuse or confound study treatments or assessments.
23. Study center personnel, close relatives of the study center personnel (e.g., parents, children, siblings, or spouse), employees or close relatives of employees at the Sponsor company.
24. Participation in any other interventional clinical study within 30 days before treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Responder Rate on a Temple Hollowing Scale | 6 months
  A treatment responder is defined as a participant with at least a one-grade improvement from baseline on both temples concurrently on the Galderma Temple Volume Deficit Scale (GTVDS, a 4-grade scale rangings are none (0), mild (1), moderate (2), severe (3) temple hollowing) as assessed by the Blinded Evaluator at 6 months after last treatment for the Treatment group and 6 months after baseline for the Control group.

SECONDARY OUTCOMES:
Responder Rate on a Temple Hollowing Scale | 3, 9 and 12 months
  A treatment responder is defined as a participant with at least a one-grade improvement from baseline on both temples concurrently on the Galderma Temple Volume Deficit Scale (GTVDS, a 4-grade scale rangings are none (0), mild (1), moderate (2), severe (3) temple hollowing). Assessed by Blinded Evaluator at 3, 9 and 12 months after last treatment for the Treatment group and at 3 months after baseline for the Control group.
Proportion of Participants Improved | 3, 6, 9 and 12 months
  Proportion of participants, defined by having at least "improved" (improved, much improved or very much improved) on the Global Aesthetic Improvement Scale (GAIS, with ratings are "Very much improved", "Much improved", "Improved", "No change" and "Worse"), on both sides of the face (each temple) concurrently, as assessed by the participant and the Treating Investigator, respectively, at 3, 6, 9 and 12 months after last treatment for the Treatment group.
Proportion of Participants Improved | 3 and 6 months
  Proportion of participants, defined by having at least "improved" (improved, much improved or very much improved) on the GAIS (with ratings are "Very much improved", "Much improved", "Improved", "No change" and "Worse"), on both sides of the face (each temple) concurrently, as assessed by the participant and the Treating Investigator, respectively, at 3 and 6 months after optional treatment for the no-treatment Control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Galderma Investigational Site #6340, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No